CLINICAL TRIAL: NCT06104865
Title: Sound Therapy for Adults With Chronic Tinnitus, Using ((Resound Tinnitus Relief)) Mobile Application, in Qatar, 2023.
Brief Title: Tinnitus Sound Therapy Using Mobile Application.
Acronym: TST
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Basel Samman (Other Government)
Collaborators: Primary Health Care Corporation, Qatar (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Basel Samman, Otolaryngology Cosultant, Primary Health Care Corporation, Qatar
Organization: Primary Health Care Corporation, Qatar (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: phc56325
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Tinnitus
Keywords: Tinnitus; Chronic Tinnitus; Adults; Sound Therapy; Mobile Application; Relieve; Relief; Resound
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Intervention Model Description: Single arm clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tinnitus Sound Therapy (Experimental): Resound Tinnitus Application, different sounds will be presented over a six months period of time on the speaker of the mobile handset in the background for 30 mins twice a day at least, loudness near but less than the tinnitus intensity itself.
  Interventions: Behavioral: Tinnitus Sound Therapy using (Resound Tinnitus relief) mobile application

INTERVENTIONS:
Behavioral: Tinnitus Sound Therapy using (Resound Tinnitus relief) mobile application — Patient exposure to relieving sound(wind, rain, ocean waves, etc) of his own choice from the mobile phone application and using this effect with time to accommodate the brain to neglect the negative effects of tinnitus.

SUMMARY:
Over the years Tinnitus Sound Therapy (TST) has been undergoing rigorous modification according to the availability of various technologies such as Hearing Aids, personal amplification devices, mp3 players, and now mobile phones. Now more than ever, it is a great opportunity to enhance accessibility, flexibility and engagement of TST as it is easy to personalize, provide tailored therapy program as well as obtaining feedback and real-time monitoring allows us to record progress of the program while keeping the cost low, which benefits to avoid purchasing personal amplification device or Hearing Aids, and hence allowing large number of people to access the service to improve the quality of life affected by Tinnitus.

The offers by mobile phone applications are too huge to avoid as the interface has gaming elements, progress tracking, reminders, and support networks, therefore providing enjoyable experience. Integration of various multimodalities into a single platform including sound therapy, relaxation exercises and educational resources addresses both the auditory and psychological aspects of tinnitus.

Our study focuses on personalized sound therapy. Real-time monitoring of progress and the effectiveness of such research will show potential to revolutionize the delivery of TST conveniently as a routine treatment for the patients that fit the inclusion criteria.

DETAILED DESCRIPTION:
Tinnitus is the sound perception of ((ringing, hissing, buzzing, etc.)), in the absence of an external stimulus. If persistent and intolerable or sufficiently bothersome, tinnitus can cause functional impairment in thought processing, emotions, hearing, sleep, and concentration, all of which can affect quality of life. The negative effect on quality of life due to chronic tinnitus has been reported to adversely affect all 5 measures of validated health related quality of life surveys including mobility, self-care, performance of usual activities, pain and/or discomfort, and anxiety/depression.

The prevalence of tinnitus ranges from 8% to 25.3% of the US population whereas in other nations similarly prevalence ranges from 4.6% to 30%. The severity of tinnitus is higher with increasing age and is more prevalent in men (10.5%) than in women (8.8%). In some populations, it's even more prevalent than back and neck pain, knee problems and diabetes milletus.

The management of Tinnitus is difficult and usually fails with the variety of treatment modality, as yet no drug has been approved for tinnitus by a regulatory body (e.g. the European Medicines Agency or US Food and Drug Administration), hens there is a need for a method that gathers the cognitive and behavioral therapy to relieve the Tinnitus, and this is where the Tinnitus Sound Therapy fits in.

The American Academy of Otolaryngology - Head and Neck Surgery Foundation (AAO-HNSF) published its multidisciplinary, evidence-based practice guidelines for the management of tinnitus, a briefing of the AAO-HNSF recommendations regarding Tinnitus treatment options:

Clinicians should not routinely recommend medications like antidepressants, anticonvulsants, anxiolytics, or intratympanic medications for a primary indication of treating persistent, bothersome tinnitus, Clinicians should not recommend dietary supplements like Ginkgo biloba, melatonin, zinc … for treating patients with persistent, bothersome tinnitus, no recommendation can be made regarding the effect of acupuncture in patients with persistent bothersome tinnitus, Clinicians should not recommend transcranial magnetic stimulation for the routine treatment of patients with persistent, bothersome tinnitus, Clinicians should recommend a hearing aid evaluation for patients with hearing loss and persistent, bothersome tinnitus, Clinicians may recommend sound therapy and cognitive behavioral therapy to patients with persistent bothersome tinnitus.

Sound therapy is the use of an instrument (Hearing Aid, Mobile, Laptop …) to generate a sound that the patient will hear as a back ground during the daily life activities, for a certain time on a daily basis for the period of several months, this sound volume is set to be just less than the patient's own tinnitus. The nature of this sound can be a wide band noise (white noise), a variety of nature sounds (River, waterfall, Wind, Birds …), music, etc. The aim is to distract and habituate the patient from focusing on his tinnitus and enable him/her to focus more on the daily life activities so that the tinnitus will no longer be an obstacle preventing the patient from enjoying life.

Modalities of Sound Therapy generators include:

Environmental enrichment devices (Tabletop sound machines generate, CD recordings or personal audio players generate music, speakers, Fans, TV, radio, Smartphones, or tablets with apps specifically created to produce a variety of sounds that aid in tinnitus relief). Hearing aids (Digital signal processing devices allow for flexibility in manipulating the acoustic signal based on the patient's hearing loss severity and audiometric configuration promoting a (masking/partial masking effect), Sound generators (Ear-level sound generators that produce broadband noise(s) (eg, white noise, pink noise) are a choice for patients with normal or near-normal audiometric thresholds, available in in-the-ear or behind-the-ear styles), Combination tinnitus instruments (Contain hearing aid circuit and noise-producing circuit in the same device may be connected by Bluetooth to any device like Laptops or Mobiles).

Our aim in the study is to use the Mobile, with a specific application (RESOUND TINNITUS RELIEF), to generate the treatment sound, this application has a variety of nature sounds (Birds, Bubbles, Crickets, Brook, Fire, Rain, Waves, Wind …), so the patient will choose the sound, which is most relieving one for him, to be used as his own specific treating sound. The patient will listen to this sound and keep it as a background for at least 60 min per day, for a period of 6 months daily. The same application (RESOUND TINNITUS RELIEF) was used for a Sound Therapy in a previous research.

In recent years, many applications on mobile phones have been developed and introduced to perform calming or masking effects for tinnitus patients.

Many studies published so far related to conventional sound therapy using an external device such as an amplification device or tinnitus masker reports to reduce the effect of tinnitus. Kim et al, (2014), used Mp3 player to provide sound therapy with different stimuli such as Narrow Band Noise (NBN), Wide Band Noise (WBN) and mixed Noise and reported improvement on Tinnitus Handicap Inventory (THI) and visual-analogue scale (VAS) values. Additionally in a study, Suziki et al. (2016) reported that there was reduction in the THI values when individual customized approach was used. However, in a review conducted by Sereda et al. (2018) showed that one type of device was not better than the other type. Alam et al (2017), in a study reported that the presentation of masking stimuli using mobiles for 6 months had a significant success in reducing the severity of tinnitus and improvement in quality of life. A recent study done by Kutyba et al. (2021) reports a decrease in tinnitus symptoms measured by THI and TFI both when a continuous use of sound therapy for 6 months was presented through a mobile application (RESOUND TINNITUS RELIEF). To further conclude, the same Kutyba et al(2022) continued the study and reported to achieve lower negative emotions and reduced overall tinnitus severity. The Tinnitus progress during the sound treatment was evaluated by two inventory questionnaires, Tinnitus Handicap Inventory (THI) and visual-analogue scale (VAS), these two questionnaires aim to study the Patient's sensation of his own tinnitus and the psychological effect of tinnitus on the patient's daily life activities (DLA), before, During (after 3 months of the start of study), and after the end of the Sound Treatment.

Even though significant data is available from these and many other researches, there is a lack of objective measurement of time the mobile apps were used by the patients at home in all the studies, there was also lack of information of usage of other forms of treatment during the researched.

Our study aims to evaluate effectiveness of mobile app alone (RESOUND TINNITUS RELIEF), to provide sound therapy for Tinnitus patients, and then evaluate the treatment results by using the THI and the VAS tinnitus evaluation questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* - Adults.
* Chronic tinnitus for more than 6 months.
* Subjective tinnitus.
* Tinnitus affecting quality of life, limiting daily life activities, and causing distress.
* Physically and mentally fit and able to fill in the questionnaires themselves.
* Persons who have a mobile phone with Android or iOS.

Exclusion Criteria:

* - Intermittent tinnitus.
* Tinnitus not affecting quality of life, not limiting daily life activities, and not causing distress.
* Objective tinnitus.
* Severe or profound hearing loss.
* No device enabling the use of the application (Patient has no mobile phone).
* Vulnerable group of patients (Pregnant women, Patients with physical or mental disabilities, Patients older than 65 years, Children under 18 years, Prisoners, Refugees)
* Patients with physical disabilities that prevent the patients from using the mobile.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Measure the severity of Chronic tinnitus after intervention using THI scale of tinnitus measurement | 6 months
  Tinnitus Handicap Inventory (THI) is a Self-reporting measure of the impact of tinnitus on the daily life. Three subscales: functional, emotional and catastrophic reactions. The participant will choose yes, sometimes, and no. A maximum of 100 can be scored and the greater the score, the greater the severity. An improvement of at least 20 points or more reflects clinically important change in the severity of tinnitus.

SECONDARY OUTCOMES:
Measure the severity of Chronic tinnitus after intervention using VAS scale of tinnitus measurement | 6 months
  The visual analog scale (VAS) is a validated, subjective measure of Tinnitus. Scores are recorded by making a handwritten mark on a 10-cm line scale that represents a continuum between "no tinnitus = score 0" and "worst tinnitus = score 10.".

CONTACTS AND LOCATIONS:
Overall Officials: Basel M Samman, Doctor, Principal Investigator — Ministry of Public Health Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: - Effect of Different Sounds on the Treatment Outcome of Tinnitus Retraining Therapy Bong Jik Kim,1,2 Sung-Won Chung,1 Jae Yun Jung,1 and Myung-Whan Suhcorresponding author, Clin Exp Otorhinolaryngol. 2014 Jun; 7(2): 87-93. Published online 2014 May 21. — https://pubmed.ncbi.nlm.nih.gov/24917903/
- See also: Effectiveness of sound therapy in patients with tinnitus resistant to previous treatments: importance of adjustments, Flavia Alencar de Barros Suzuki, Fabio Akira Suzuki, Fernando Kaoru Yonamine, Ektor Tsuneo Onishi, Norma Oliveira Penido, PMID: 26541232 — https://pubmed.ncbi.nlm.nih.gov/26541232/
- See also: Sound therapy (using amplification devices and/or sound generators) for tinnitus in adults Magdalena Sereda,corresponding author Jun Xia, Amr El Refaie, Deborah A Hall, and Derek J Hoare, Cochrane Database Syst Rev. 2018 Aug; 2018(8): CD013094. Publishe — https://pubmed.ncbi.nlm.nih.gov/30589445/
- See also: Efficacy of TRT Using Noise Presentation from Mobile Phone Md. Noorain Alam, Manish Gupta, Sanjay Munjal & Naresh K. Panda, Indian Journal of Otolaryngology and Head & Neck Surgery volume 69, pages 333-337 (2017)Cite this article, — https://link.springer.com/article/10.1007/s12070-017-1141-2
- See also: Effectiveness of tinnitus therapy using a mobile application, Eur Arch Otorhinolaryngol. 2022; 279(3): 1257-1267. Published online 2021 Mar 30. , Justyna Kutyba,corresponding author1 Elżbieta Gos,1 Wiesław Wiktor Jędrzejczak — https://link.springer.com/article/10.1007/s00405-021-06767-9
- See also: American Tinnitus Association, Tinnitus Handicap Inventory (THI; Newman et al., 1996), — https://novopsych.com.au/assessments/diagnosis/tinnitus-handicap-inventory-thi/
- See also: Visual Analogue Scales as a Tool for Initial Assessment of Tinnitus Severity: Psychometric Evaluation in a Clinical Population, Danuta Raj-Koziak, Elzbieta Gos, Weronika Swierniak, Joanna J Rajchel, Lucyna Karpiesz, Iwona Niedzialek, Elzbieta Wlodarczyk, — https://pubmed.ncbi.nlm.nih.gov/30439712/